CLINICAL TRIAL: NCT03723356
Title: Linking Cognitive Functioning to Multimodal Imaging in Multiple Sclerosis
Brief Title: Linking Cognitive Functioning to Multimodal Imaging in Multiple Sclerosis (MS)
Status: Terminated | Type: Observational
Why Stopped: due to low enrollment
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 17-00238
Record Dates: First submitted 2018-09-27; First posted 2018-10-29 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Multiple Sclerosis; Cognition Disorders
MeSH Terms: conditions — Multiple Sclerosis; Cognition Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MS Patients: Definite diagnosis of RRMS
  Interventions: Diagnostic Test: Siemens Biograph mMR (molecular MR); Diagnostic Test: fMRI; Diagnostic Test: Diffusion Spectrum Imaging (DSI)
- Healthy Controls: gender aged match healthy
  Interventions: Diagnostic Test: Siemens Biograph mMR (molecular MR); Diagnostic Test: fMRI; Diagnostic Test: Diffusion Spectrum Imaging (DSI)

INTERVENTIONS:
Diagnostic Test: Siemens Biograph mMR (molecular MR) — 5mCi of the radiotracer FDG administered intravenously as a bolus over 30s. After injection, emission data will be collected for 60 min,
Diagnostic Test: fMRI — High-resolution T1-weighted structural image will be acquired using an MP2RAGE sequence. Subject will beasked to look at the cross hair on a screen andnot fixate on any one thought.
Diagnostic Test: Diffusion Spectrum Imaging (DSI) — DSI allows for more accurate characterization of diffusion,overcomes traditional dMRI artifacts, and is capable of more precise and detailedcharacterization of white matter fibers

SUMMARY:
Multiple sclerosis (MS) is the most common progressive neurologic disorder to occur in adults of working-age. Despite longstanding recognition of cognitive impairment as a symptom of MS, two obstacles in measurement have limited understanding its biological basis, and therefore identifying targeted options for management. First is the absence of a sensitive and precise measure of cognitive impairment. Second is the absence of an index of disease status linked to brain pathophysiology and cognitive performance. This project overcomes both obstacles to link cognitive impairment to MS disease biomarkers. The absence of a sensitive and precise measure of cognitive impairment, along with the absence of an index of disease status linked to brain pathophysiology and cognitive performance, limits the understanding of the biological basis for multiple sclerosis (MS). This project overcomes both obstacles to link cognitive function to MS disease biomarkers, and provides preliminary evaluation of a disease modifying therapy (Tecfidera) for preserving cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
2. Male and Female subjects between 18 and 45 years
3. WRAT-4 Reading [127] standard score > 85
4. Able to undergo neuroimaging data collection procedures. For MS Participants
5. Definite diagnosis of RRMS [128]
6. EDSS of 0 to 6.0
7. Adequate vision as as reported by the participant (with correction if applicable)
8. Clinically prescribed Tecfidera, Tysabri or Ocrevus therapy by treating neurologist, with first dose being within 3 months + 14 days from baseline visit
9. At baseline visit, concurrent medications to be kept constant over three months prior to data collection visits
10. No relapse or steroids in previous month

Exclusion Criteria:

1. Unable or unwilling to provide informed consent.
2. Beck Depression Inventory-Fast Screen (BDI-FS) [129, 130] score of 4 or more
3. Current alcohol or other substance use disorder
4. Primary psychiatric disorder that would adversely influence ability to participate
5. Other neurological condition associated with cognitive impairment (e.g., epilepsy, brain injury)
6. Other serious uncontrolled medical condition (e.g., cancer or acute myocardial infarction)
7. Learned English language after 12 years of age
8. For low absolute low lymphocyte count (ALC), USPI guidance will be utilized.

   For MS participants:
9. Lemtrada, Cladribine, Mitoxantrone

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 20 MS participants and 10 healthy controls. However, the data analysis is planned for 15 MS participants and 10 healthy control participants. It is expected that 15 MS subjects and 10 healthy controls will complete 12 months.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-01-09 (Actual); Study Completion 2021-01-09 (Actual)

PRIMARY OUTCOMES:
intraindividual variation (ie IIV) in reaction times across the trials of the Attention Network Test (ANT) | Baseline
  Attention Network Test (ANT) is a cognitive reaction time test administered on the computer, where the subject indicates when they see a target on a screen.
intraindividual variation (ie IIV) in reaction times across the trials of the Attention Network Test (ANT) | 3 Months
  Attention Network Test (ANT) is a cognitive reaction time test administered on the computer, where the subject indicates when they see a target on a screen.
intraindividual variation (ie IIV) in reaction times across the trials of the Attention Network Test (ANT) | 6 Months
  Attention Network Test (ANT) is a cognitive reaction time test administered on the computer, where the subject indicates when they see a target on a screen.
intraindividual variation (ie IIV) in reaction times across the trials of the Attention Network Test (ANT) | 9 Months
  Attention Network Test (ANT) is a cognitive reaction time test administered on the computer, where the subject indicates when they see a target on a screen.
intraindividual variation (ie IIV) in reaction times across the trials of the Attention Network Test (ANT) | 12 Months
  Attention Network Test (ANT) is a cognitive reaction time test administered on the computer, where the subject indicates when they see a target on a screen.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.